CLINICAL TRIAL: NCT00729014
Title: A Study of Drug-Induced Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Responsible Party: Fe-Lin L Wu, Ph.D., Director, National Taiwan University Hospital
Other Study IDs: 200804062R
Record Dates: First submitted 2008-08-01; First posted 2008-08-06 (Estimated); Last update posted 2008-08-06 (Estimated); Status verified 2008-05

CONDITIONS: End Stage Renal Disease
Keywords: herbal nephropathy; Chinese herbal nephropathy; nephrotoxicity; renal disease; adverse drug reaction; Chinese herbal medicine
MeSH Terms: conditions — Kidney Failure, Chronic; Kidney Diseases; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to identify incidence of Chinese herb nephropathy in a medical center

DETAILED DESCRIPTION:
This is a retrospective study, by computer screening, chart review and phone survey to find herbal nephropathy and determine the cause-relationship.

Using ICD-9-CM code as a tool to screen the newly diagnosed ESRD in NTUH computer data base, and divided patients into those with underlying disease(s) that cause the renal failure and those without.

ELIGIBILITY:
Inclusion Criteria:

* patient who was newly diagnosed as end stage renal disease who need dialysis

Exclusion Criteria:

* started dialysis before 2000

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: a medical center
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2008-05; Primary Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
The incidence of herbal nephropathy | 5 years

SECONDARY OUTCOMES:
The epidemiology of primary diagnosis for end stage renal disease in Taiwan | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kwan-Dun Wu, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan